CLINICAL TRIAL: NCT01855139
Title: Belgian Real Life Non-interventional Study (NIS) on Xarelto® in Non-valvular Atrial Fibrillation (AF) Patients Treated for the Prevention of Stroke and Systemic Embolism (BOX-AF)
Brief Title: Belgian Real Life Non-interventional Study (NIS) on Xarelto in Non-valvular Atrial Fibrillation (AF) Patients Treated for the Prevention of Stroke and Systemic Embolism
Acronym: BOX-AF
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16851; XA1313BE (Other: Company internal)
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation; Stroke; Systemic embolism; Oral anticoagulation; Real-life setting; Preventive measure
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rivaroxaban
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — 15 mg OD or 20 mg OD

SUMMARY:
The objective of this NIS is to assess in a real-life setting, usage patterns and associated outcomes in the management (healthcare resource utilisation and associated costs) of patients with non-valvular AF treated with Xarelto, in accordance with the terms of the European marketing authorization and the Belgian reimbursement criteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old with a confirmed diagnosis of non-valvular atrial fibrillation
* Patients must in addition present with at least one of following risk factors:

  * prior stroke, TIA (transient ischemic attack) or non-CNS (central nervous system) systemic embolism
  * left ventricular ejection fraction of < 40%
  * symptomatic heart failure, New York Heart Association class 2 or higher
  * age ≥75 years
  * age ≥65 years in combination with either diabetes, coronary disease or arterial hypertension

Exclusion Criteria:

* Patients who do not fulfil the Belgian reimbursement criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory or hospitalized patients coming from the cardiology clinic of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with major bleedings | 1 year or 30 days after end of rivaroxaban
Number of patients with symptomatic thromboembolic events | 1 year or 30 days after end of rivaroxaban
All-cause mortality | 1 year or 30 days after end of rivaroxaban
Adverse events | 1 year or 30 days after end of rivaroxaban
Treatment satisfaction measured by means of Anti-clot treatment scale (ACTS) | 1 year or 30 days after end of rivaroxaban
Quantities of resource use consumption | 1 year or 30 days after end of rivaroxaban

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Belgium